CLINICAL TRIAL: NCT01407601
Title: Food Supplementation With Vitamin K2 to Activate MGP as an Endogenous Inhibitor of Vascular Calcification in Hemodialysis Patients
Brief Title: Vitamin K2 Supplementation to Activate Matrix Gla Protein (MGP) as Endogenous Inhibitor of Vascular Calcification in Hemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: CTC Aachen, University Hospital of the RWTH Aachen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: EK 111/07
Record Dates: First submitted 2011-07-29; First posted 2011-08-02 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-08

CONDITIONS: CKD 5D, Hemodialysis
Keywords: vitamin K; MK-7; Hemodialysis; vascular calcification; Matrix Gla protein; Osteocalcin
MeSH Terms: conditions — Vascular Calcification

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 45 µg MK-7 (Experimental): 45 µg MK-7 daily over 6 weeks
  Interventions: Dietary Supplement: daily supplementation of MK-7 over 6 weeks
- 135 µg MK-7 (Experimental): 135 µg MK-7 daily over 6 weeks
  Interventions: Dietary Supplement: daily supplementation of MK-7 over 6 weeks
- 360 µg MK-7 (Experimental): 360 µg MK-7 daily over 6 weeks
  Interventions: Dietary Supplement: daily supplementation of MK-7 over 6 weeks

INTERVENTIONS:
Dietary Supplement: daily supplementation of MK-7 over 6 weeks — once daily intake of MK-7 prior to dialysis over 6 weeks

SUMMARY:
Vascular calcification (VC) is a predictor of cardiovascular morbidity and mortality. Hemodialysis (HD) patients suffer from severe vascular calcifications. Matrix Gla protein (MGP) is a central calcification inhibitor of the arterial wall and its activity depends on vitamin K-dependent γ-glutamate carboxylation. Noncarboxylated MGP, formed as a result of vitamin K deficiency, is associated with cardiovascular disease. Recent studies pointed towards poor vitamin K status in HD patients. We therefore aim to investigate whether daily vitamin K2 (MK-7) supplementation improves the bioactivity of vitamin K-dependent proteins in HD patients as assessed by circulating dephospho-noncarboxylated MGP (dp-ucMGP), noncarboxylated osteocalcin (ucOC) and noncarboxylated prothrombin (ucFII; PIVKA-II).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* minimum of 3 months of hemodialysis
* written consent

Exclusion Criteria:

* chronic or acute bowel disease
* soy bean allergy
* active Vitamin K Supplementation
* oral anticoagulation with vitamin K Antagonists (coumarins)
* systemic therapy using steroids
* positive history for thrombosis or embolism
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Reduction of plasma levels of noncarboxylated MGP | after 6 weeks of supplementation
  Noncarboxylated MGP levels [pmol/L] will be determined from plasma samples by a non-commercial ELISA. Plasma samples will be obtained each week of the six-week treatment period and compared to baseline values.
Reduction of plasma levels of noncarboxylated osteocalcin | after 6 weeks of supplementation
  Noncarboxylated osteocalcin levels [ng/ml] will be determined from plasma samples by a commercial ELISA. Plasma samples will be obtained each week of the six-week treatment period and compared to baseline values.
Reduction of plasma levels of inactive prothrombin (PIVKA-II) | after 6 weeks of supplementation
  PIVKA-II levels [ng/ml] will be determined from plasma samples by a commercial ELISA. Plasma levels at the end of the six-week treatment period will be compared to baseline levels.

SECONDARY OUTCOMES:
increase of plasma levels of carboxylated MGP | after 6 weeks of supplementation
  Carboxylated MGP levels [pmol/L] will be determined from plasma samples by a non-commercial ELISA. Plasma samples will be obtained each week of the six-week treatment period and compared to baseline values.
increase of plasma levels of carboxylated osteocalcin | after 6 weeks of supplementation
  Carboxylated MGP levels [ng/ml] will be determined from plasma samples by a commercial ELISA. Plasma samples will be obtained each week of the six-week treatment period and compared to baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Westenfeld, MD, Principal Investigator — University Clinic of the RWTH Aachen; Georg Schlieper, MD, Study Chair — University Clinic of the RWTH Aachen; Stefan Holzmann, MD, Study Chair — Dialysis Unit Erkelenz, Germany; Stephan Heidenreich, MD, Study Chair — KfH Dialysis Centre Aachen, Schurzelter Strasse; Juergen Floege, MD, Study Director — University Clinic of the RWTH Aachen; Thilo Krueger, MD, Study Chair — University Hospital of the RWTH Aachen
Locations (3):
- Germany (3):
  - KfH Dialysis Unit Aachen, Aachen, North Rhine-Westphalia
  - University Hospital of the RWTH Aachen, Aachen, North Rhine-Westphalia
  - Dialysis Unit Erkelenz, Erkelenz, North Rhine-Westphalia

REFERENCES:
- [Derived] Westenfeld R, Krueger T, Schlieper G, Cranenburg EC, Magdeleyns EJ, Heidenreich S, Holzmann S, Vermeer C, Jahnen-Dechent W, Ketteler M, Floege J, Schurgers LJ. Effect of vitamin K2 supplementation on functional vitamin K deficiency in hemodialysis patients: a randomized trial. Am J Kidney Dis. 2012 Feb;59(2):186-95. doi: 10.1053/j.ajkd.2011.10.041. Epub 2011 Dec 9. PMID 22169620